CLINICAL TRIAL: NCT06998186
Title: The Effect Of Discharge Education And Telephone Counseling in Pediatric Cardiac Surgery Patients
Brief Title: Discharge Education And Telephone Counseling in Pediatric Cardiac Surgery Patients
Acronym: telcon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: telcounseling
Record Dates: First submitted 2024-09-18; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Anxiety; Stress; Quality of Life; Counselling
Keywords: pediatric; surgery; telephone counselling; discharge; stress; quality of life
MeSH Terms: conditions — Cardiovascular Diseases; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): standard care. No telephone counselling.
- Discharge Education And Telephone Counseling (Experimental): Discharge and instruction on medication usage Providing training on discharge education to parents of cardiac surgery patients (10-15 minutes on average) (using educational materials on discharge and medications)
  Interventions: Behavioral: Discharge Education And Telephone Counseling

INTERVENTIONS:
Behavioral: Discharge Education And Telephone Counseling — Providing training on discharge education to parents of cardiac surgery patients.
  Providing telephone counseling for 6 months
  Arms: Discharge Education And Telephone Counseling

SUMMARY:
It was aimed to evaluate the effect of discharge education and telephone counselling applied to parents of 0-6 years old pediatric cardiac surgery patients on postoperative patient outcomes, quality of life, anxiety, and stress levels of parents.

DETAILED DESCRIPTION:
H0: Discharge education and telephone counselling applied to parents of paediatric cardiac surgery patients has no effect on postoperative patient outcomes (weight gain, tachypnoea/cyanosis/chest pain, increase in activity, complication status), parents' anxiety, stress and quality of life.

H1: Discharge education and telephone counselling applied to parents of paediatric cardiac surgery patients have an effect on postoperative patient outcomes (weight gain, tachypnoea/cyanosis/chest pain, increase in activity, complication status), parents' anxiety, stress and quality of life.

Data Collection:

After the child and his family are informed about the study, their written informed consent will be obtained. According to the randomisation scheme, patients will be divided into experimental and control groups by stratified randomisation method.

The parents of the patients in the study group will get pre-discharge education. The clinic's routine will continue for the children in the control group, and they won't receive any training. The researcher will conduct a telephone consultation to assess the outcomes of the patients in both groups, as well as the parents' quality of life, anxiety, and stress levels.

ELIGIBILITY:
Inclusion Criteria:

* The child's age ranges from 0 to 6 years old.
* Possessing congenital heart disease
* Planning for pediatric heart surgery
* Receiving inpatient care;
* Receiving a recent diagnosis and beginning therapy
* The parent willingly consents to participate in the study;
* There isn't another child in the family who has CHD.
* Getting the parent's consent on paper

Exclusion Criteria:

* Suffering from another illness
* The child is nearing the end of their life.
* The child and family have expressed a lack of willingness to engage in the study.
* Illiteracy of the parents
* The child and family do not know Turkish

Ages: 60 Days to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
anxiety with State-Trait Anxiety Inventory | change in the State-Trait Anxiety Inventory (baseline-at hospital, 1st, 3rd and 6th months after the discharge) ]
  Anxiety assessment with State-Trait Anxiety Inventory by parent
quality of life with World Health Organization Quality of Life Scale Short Form Turkish Version | change in the World Health Organization Quality of Life Scale Short Form Turkish Version (WHOQOL-BREF-TR) (baseline-at hospital, 1st, 3rd and 6th months after the discharge) ]
  quality of life with World Health Organization Quality of Life Scale Short Form Turkish Version (WHOQOL-BREF-TR)
stress with Parental Stress Scale-Short Form | change in the Parental Stress Scale (baseline-at hospital, 1st, 3rd and 6th months after the discharge)
  Stress assessment with Parental Stress Scale-Short Form by parent

SECONDARY OUTCOMES:
Post-Surgery Patient Outcomes | 1st, 3rd and 6th months after the discharge
  change in health status, physical problems, physical symptoms, if any, adaptation to normal life, problems experienced, etc. besides regarding nutrition, breastfeeding, weight gain, oxygen saturation, pulse, respiration, pain, cleaning/bathing, wound healing, presence of infection, neurodevelopmental and motor behaviors, activity level, and medications after the discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Gulcin Ozalp Gerçeker, Assoc. Prof., Principal Investigator — Dokuz Eylul University
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No